CLINICAL TRIAL: NCT02260531
Title: A Phase II Study of Cabozantinib Alone or in Combination With Trastuzumab in Breast Cancer Patients With Brain Metastases
Brief Title: Cabozantinib +/- Trastuzumab In Breast Cancer Patients w/ Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Exelixis (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-359
Record Dates: First submitted 2014-09-17; First posted 2014-10-09 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Brain Tumor - Metastatic
Keywords: Metastatic breast cancer and brain metastases; HER-2 Positive Breast Cancer; ER-Positive PR-Positive HER-2 Negative Breast Cancer; ER-Negative PR-Negative HER2-Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Triple Negative Breast Neoplasms | interventions — cabozantinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 - Cabozantinib, Trastuzumab for HER2+ (Experimental): HER2-positive
  * Cabozantinib- orally administered daily per treatment cycle, 60 mg per day
  * Trastuzumab- IV administered once per cycle, 8 mg/kg IV loading dose followed by 6 mg/kg IV Cycle duration equals 3 weeks. Patients are treated indefinitely based on unacceptable toxicity, disease progression, or withdrawal for other reasons.
  Interventions: Drug: Cabozantinib; Drug: Trastuzumab
- Cohort 2 - Cabozantinib for ER+ and/or PR+ (Experimental): Hormone receptor-positive (ER+ and/or PR+)
  - Cabozantinib- orally administered daily per treatment cycle, 60 mg per day Cycle duration equals 3 weeks. Patients are treated indefinitely based on unacceptable toxicity, disease progression, or withdrawal for other reasons.
  Interventions: Drug: Cabozantinib
- Cohort 3 - Cabozantinib for ER-, PR-, HER2- (Experimental): Triple negative (ER-, PR-, HER2-)
  - Cabozantinib- orally administered daily per treatment cycle, 60 mg per day Cycle duration equals 3 weeks. Patients are treated indefinitely based on unacceptable toxicity, disease progression, or withdrawal for other reasons.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib
  Other Names: Cometriq®
Drug: Trastuzumab
  Other Names: Herceptin
  Arms: Cohort 1 - Cabozantinib, Trastuzumab for HER2+

SUMMARY:
This research study is evaluating the effectiveness of the drug called cabozantinib (alone or in combination with trastuzumab) as a possible treatment for advanced breast cancer in which the cancer has spread to the brain.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved cabozantinib for your specific disease but it has been approved for other uses.

Few treatments exist for brain metastases from breast cancer. Radiation and surgery are generally included as a possible standard of care treatments for this diagnosis.

In this research study, the investigator are looking at how well cabozantinib works in treating breast cancer that has spread to the brain. Cabozantinib has been used in some phase I studies and information from those other research studies suggests that cabozantinib may help to shrink or stabilize the participant's breast cancer. In addition, information from these studies has shown that cabozantinib may pass through the blood brain barrier (a protective layer that prevents most large molecules and cells found in the blood from entering the brain tissue) and may be an effective treatment for brain metastases.

If the participant has HER2-positive breast cancer, they will receive trastuzumab in addition to cabozantinib. Trastuzumab is an FDA approved drug for the treatment of HER2-positive metastatic breast cancer. However, the combination of cabozantinib and trastuzumab has not yet been tested. Trastuzumab may help to shrink or stabilize breast cancer in combination with cabozantinib. If the participant's breast cancer is HER2-negative, they will not receive trastuzumab as part of this clinical trial.

The names of the study interventions involved in this study are:

* Cabozantinib (XL184)
* Trastuzumab (herceptin) (participants with HER2-positive disease only)

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast cancer, with stage IV disease.
* New or progressive CNS lesions, as assessed by the patient's treating physician.
* For patients who have received prior cranial radiation, no increase in corticosteroid dose in the week prior to the baseline brain MRI
* Discontinued prior therapy (with the exception of trastuzumab for patients with HER2+ breast cancer)
* Recovery to baseline or ≤ Grade 1 CTCAE v.4.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy;
* The subject has an ECOG performance status of 0 or 1
* Patients must have normal organ and marrow function and laboratory values as follows within 14 days before the first dose of cabozantinib
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s)
* Subjects of childbearing potential must not be pregnant at screening.
* Patients on bisphosphonates may continue receiving bisphosphonate therapy during study. Patients wanting to initiate bisphosphonate therapy may do so.
* The subject has had an assessment of all known disease sites eg, by computerized tomography (CT) scan, magnetic resonance imaging (MRI), bone scan as appropriate, within 28 days before the first dose of cabozantinib

Exclusion Criteria:

* The subject has received cabozantinib or another c-Met inhibitor (please note ARQ 197 is not considered a MET inhibitor for purposes of this study given data to suggest it inhibits tubulin)
* The subject has uncontrolled, significant intercurrent or recent illness
* Leptomeningeal disease as the only site of CNS involvement
* Known contraindication to MRI with gadolinium contrast, such as cardiac pacemaker, shrapnel, or ocular foreign body
* More than 2 seizures over the last 4 weeks prior to study entry
* Grade 1 or higher CNS hemorrhage on baseline brain MRI, or history of grade 2 or higher CNS hemorrhage within 12 months
* Has experienced clinically-significant GI bleeding within 6 months before first dose of cabozantinib; hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood within 3 months before the first dose of cabozantinib; any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of cabozantinib
* The subject has tumor in contact with, invading or encasing any major blood vessels
* The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants. Low dose aspirin (≤ 81 mg/day), low-dose warfarin ( ≤1 mg/day), and prophylactic LMWH are permitted.
* The subject has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥1.3 × the laboratory ULN within 7 days before the first dose of cabozantinib.
* Inability to swallow intact tablets
* Pregnant or lactating females
* Diagnosis of another malignancy within 2 years before the first dose of cabozantinib, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy
* Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* The subject is known to be positive for the human immunodeficiency virus (HIV)
* Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* QTcF > 500 msec on average of screening EKGs performed within 28 days of first dose of cabozantinib. Three EKGs must be performed at screening. If the average of these three consecutive results for QTcF is > 500 msec, the subject is ineligible.
* Active infection requiring IV antibiotics at Day 1 of cycle 1
* No prior lapatinib within 7 days prior to initiation of protocol treatment
* Receive concurrent investigational agents while on study
* Receive any concurrent chemotherapy, radiotherapy, or hormonal therapy while on study
* Previously identified allergy or hypersensitivity to components of the cabozantinib formulations
* The subject requires chronic concomitant treatment with strong CYP3A4 inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Leone JP, Duda DG, Hu J, Barry WT, Trippa L, Gerstner ER, Jain RK, Tan S, Lawler E, Winer EP, Lin NU, Tolaney SM. A phase II study of cabozantinib alone or in combination with trastuzumab in breast cancer patients with brain metastases. Breast Cancer Res Treat. 2020 Jan;179(1):113-123. doi: 10.1007/s10549-019-05445-z. Epub 2019 Sep 20. PMID 31541381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 patients were enrolled between November 2014 and June 2018
Groups:
- Cohort 1 - Cabozantinib, Trastuzumab for HER2+: HER2-positive
  * Cabozantinib- orally administered daily per treatment cycle
  * Trastuzumab- IV administered once per cycle
  * MRI- Baseline, Cycle 2 Day 1, and every 2 cycles
  * Magnetic Resonance Angiography (MRA ), Baseline, Cycle 2 Day 1,
  Cabozantinib: One, 60 mg tablet daily of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Trastuzumab: For HER2-Positive participants only. Administered by IV on day 1 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
- Cohort 2 - Cabozantinib for ER+ and/or PR+: Hormone receptor-positive (ER+ and/or PR+)
  * Cabozantinib- orally administered daily per treatment cycle
  * MRI- Baseline, Cycle 2 Day 1, and every 2 cycles
  * Magnetic Resonance Angiography (MRA ), Baseline, Cycle 2 Day 1,
  Cabozantinib: One, 60 mg tablet daily of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
- Cohort 3 - Cabozantinib for ER-, PR-, HER2-: Triple negative (ER-, PR-, HER2-)
  * Cabozantinib- orally administered daily per treatment cycle
  * MRI- Baseline, Cycle 2 Day 1, and every 2 cycles
  * Magnetic Resonance Angiography (MRA ), Baseline, Cycle 2 Day 1,
  Cabozantinib: One, 60 mg tablet daily of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
Period: Overall Study
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2-
Started | 21 | 7 | 8
Completed | 21 | 7 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2- | Total
Number analyzed (Participants) | 21 | 7 | 8 | 36
Age, Continuous [Median (Full Range); unit: years] | 52 [28 to 69] | 48 [40 to 62] | 48 [33 to 62] | 50 [28 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 7 | 8 | 36
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 19 | 5 | 8 | 32
  Race: African American | 0 | 2 | 0 | 2
  Race: More than one race | 1 | 0 | 0 | 1
  Race: Other | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 7 | 8 | 36
Prior anti-HER2 therapy-Trastuzumab [Count of Participants; unit: Participants] | 21 | 0 | 0 | 21
Prior anti-HER2 therapy-Lapatinib [Count of Participants; unit: Participants] | 10 | 0 | 0 | 10
ECOG performance status [Count of Participants; unit: Participants] — ECOG performance status:
  0 - Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  1 - Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    0 | 13 | 3 | 1 | 17
    1 | 8 | 4 | 7 | 19
Prior Stereotactic radiosurgery [Count of Participants; unit: Participants]
  Yes | 7 | 4 | 1 | 12
  No | 14 | 3 | 7 | 24
Prior Whole brain radiation [Count of Participants; unit: Participants]
  Yes | 16 | 5 | 4 | 25
  No | 5 | 2 | 4 | 11
No Prior CNS radiation [Count of Participants; unit: Participants] | 4 | 2 | 4 | 10
Surgical resection of CNS metastasis [Count of Participants; unit: Participants]
  Yes | 1 | 1 | 2 | 4
  No | 20 | 6 | 6 | 32
Sites of metastatic disease [Number; unit: participants]
  Lung | 9 | 2 | 3 | 14
  Liver | 7 | 1 | 1 | 9
  Bone | 10 | 5 | 1 | 16
  Breast (Ipsilateral or Contralateral) or chest wall | 2 | 0 | 1 | 3
  Lymph nodes | 5 | 1 | 1 | 7
Number of sites of metastases at study entry [Median (Full Range); unit: Sites] | 2 [1 to 4] | 1 [1 to 3] | 2 [1 to 3] | 2 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: CNS Objective Response Rate (ORR)
Description: The central nervous system (CNS) ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria in the evaluation CNS lesions on treatment: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease assessments occurred every 6 cycles. Patients with stable or responsive disease after completion of 6 cycles could reduce frequency of assessments to every 3 cycles. Response was evaluated up to 25 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2-
Number analyzed (Participants) | 21 | 7 | 8
percentage of participants | 5 [.2 to 24] | 14 [.4 to 58] | 0 [0 to 37]

2. Secondary Outcome: CNS Volumetric Objective Response Rate (ORR)
Description: CNS volumetric ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) defined as:
  CR
  * Complete resolution of all measurable (≥ 1 cm diameter) and non-measurable brain metastases
  * No new CNS lesions (new lesion defined as ≥ 6 mm diameter) PR
  * ≥ 50% reduction in the volumetric sum of all measurable (≥ 1 cm diameter) brain metastases compared to baseline
  * No progression of non-measurable lesions
  * No new lesions (new lesion defined as ≥ 6 mm)
  ORR also requires:
  * Stable or decreasing steroid dose
  * No new/progressive tumor-related neurologic signs or symptoms
Time Frame: Disease assessments occurred every 6 cycles. Patients with stable or responsive disease after completion of 6 cycles could reduce frequency of assessments to every 3 cycles. Response was evaluated up to 25 months .
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2-
Number analyzed (Participants) | 21 | 7 | 8
percentage of participants | 5 [0.2 to 24] | 0 [0 to 41] | 0 [0 to 37]

3. Secondary Outcome: Non-CNS Objective Response Rate (ORR)
Description: The non-central nervous system (CNS) ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria in the evaluation non-CNS lesions on treatment: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2-
Number analyzed (Participants) | 21 | 7 | 8
percentage of participants | 0 [0 to 16] | 0 [0 to 41] | 0 [0 to 37]

4. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease assessments occurred every 6 cycles. Patients with stable or responsive disease after completion could reduce frequency to every 3 cycles. In long-term follow-up, assessments occurred every 6 months until death. Follow-up time is up to 25 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2-
Number analyzed (Participants) | 21 | 7 | 8
Months | 4.1 [2.8 to 6.2] | 0.8 [0.5 to NA] — Insufficient number of participants with events | 2.4 [2.0 to NA] — Insufficient number of participants with events

5. Secondary Outcome: 12-Week Clinical Benefit Rate
Description: Clinical benefit rate (CBR) was defined as the percentage of patients achieving complete response (CR), partial response (PR), or stable disease (SD) based on RECIST 1.1 criteria by 12 weeks. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PD is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Stable disease (SD) is defined as any condition not meeting the above criteria.
Time Frame: Evaluate at 12 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2-
Number analyzed (Participants) | 21 | 7 | 8
percentage of participants | 43 [24 to 63] | 14 [0.4 to 58] | 13 [1 to 47]

6. Secondary Outcome: First Progression Site
Description: Site that a patient has his/her first tumor progression (CNS vs Non-CNS)
Time Frame: as for outcome 4
Population: Data was not collected
Groups:
- Cohort 1 - Cabozantinib, Trastuzumab for HER2+: HER2-positive
  * Cabozantinib- orally administered daily per treatment cycle, 60 mg per day
  * Trastuzumab- IV administered once per cycle, 8 mg/kg IV loading dose followed by 6 mg/kg IV Cycle duration equals 3 weeks. Patients are treated indefinitely based on unacceptable toxicity, disease progression, or withdrawal for other reasons.
  Trastuzumab
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2-
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Off-treatment patients followed every 6 months until death. Follow-up time is up to 25 months.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort 1 - Cabozantinib, Trastuzumab for HER2+: HER2-positive
  * Cabozantinib- orally administered daily per treatment cycle
  * Trastuzumab- IV administered once per cycle
  * MRI- Baseline, Cycle 2 Day 1, and every 2 cycles
  * Magnetic Resonance Angiography (MRA ), Baseline, Cycle 2 Day 1,
- Cohort 2 - Cabozantinib for ER+ and/or PR+: Hormone receptor-positive (ER+ and/or PR+)
  * Cabozantinib- orally administered daily per treatment cycle
  * MRI- Baseline, Cycle 2 Day 1, and every 2 cycles
  * Magnetic Resonance Angiography (MRA ), Baseline, Cycle 2 Day 1,
- Cohort 3 - Cabozantinib for ER-, PR-, HER2-: Triple negative (ER-, PR-, HER2-)
  * Cabozantinib- orally administered daily per treatment cycle
  * MRI- Baseline, Cycle 2 Day 1, and every 2 cycles
  * Magnetic Resonance Angiography (MRA ), Baseline, Cycle 2 Day 1,
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2-
Number analyzed (Participants) | 21 | 7 | 8
Months | 13.8 [8.2 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 5.1 [2.1 to NA] — Insufficient number of participants with events

8. Secondary Outcome: Incidence of Grade 4 Treatment-Related Toxicity
Description: All grade 4 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 4 AE of any type during the time of observation.
Time Frame: Participants should be re-evaluated for response every 6 weeks. Patients with stable or responsive disease after completion of 6 cycles may have the frequency of scans reduced to once every 3 cycles, and in long-term follow-up every 6 months until death.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2-
Number analyzed (Participants) | 21 | 7 | 8
participants | 4 [1.05 to 8.82] | 0 [0 to 2.87] | 0 [0 to 2.96]

ADVERSE EVENTS:
Time Frame: Disease assessments occurred every 6 cycles. Patients with stable or responsive disease after completion could reduce frequency to every 3 cycles. In long-term follow-up, assessments occurred every 6 months until death.
Description: All toxicities should be graded according to the Common Terminology Criteria for Adverse Events (Version 4.0)
Arm/Group | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ | Cohort 2 - Cabozantinib for ER+ and/or PR+ | Cohort 3 - Cabozantinib for ER-, PR-, HER2-
All-Cause Mortality (participants affected / at risk) | 11/21 | 3/7 | 8/8
Serious Adverse Events (participants affected / at risk) | 6/21 | 4/7 | 6/8
Other Adverse Events (participants affected / at risk) | 21/21 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ (N=21) | Cohort 2 - Cabozantinib for ER+ and/or PR+ (N=7) | Cohort 3 - Cabozantinib for ER-, PR-, HER2- (N=8)
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Lipase increased (Investigations) | 3 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Serum amylase increased (Investigations) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Cabozantinib, Trastuzumab for HER2+ (N=21) | Cohort 2 - Cabozantinib for ER+ and/or PR+ (N=7) | Cohort 3 - Cabozantinib for ER-, PR-, HER2- (N=8)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 1
Papulopustular rash (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 3 | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 2 | 1
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 0 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 0 | 1
Blurred vision (Eye disorders) | 3 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 10 | 3 | 2
Diarrhea (Gastrointestinal disorders) | 8 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 7 | 2 | 2
Nausea (Gastrointestinal disorders) | 8 | 3 | 2
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 2 | 2
Edema limbs (General disorders) | 0 | 1 | 0
Edema trunk (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 16 | 5 | 7
Gait disturbance (General disorders) | 2 | 1 | 0
Pain (General disorders) | 3 | 1 | 4
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 0 | 1
Eye infection (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 2 | 3
Alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 11 | 0 | 3
Blood bilirubin increased (Investigations) | 1 | 1 | 1
Lipase increased (Investigations) | 3 | 0 | 1
Platelet count decreased (Investigations) | 2 | 2 | 1
Serum amylase increased (Investigations) | 4 | 0 | 0
Weight loss (Investigations) | 2 | 0 | 0
Investigations - Other, specify (Investigations) | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5 | 0 | 3
Ataxia (Nervous system disorders) | 4 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 2 | 2
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 1
Sinus pain (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Confusion (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 1 | 2
Personality change (Psychiatric disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 | 2 | 2
Hot flashes (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 7 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT02260531/Prot_SAP_000.pdf